CLINICAL TRIAL: NCT05076942
Title: Groningen International Study on Sentinel Nodes in Vulvar Cancer-III, a Prospective Phase II Treatment Trial
Brief Title: Groningen International Study on Sentinel Nodes in Vulvar Cancer-III
Acronym: GROINSS-VIII
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Dutch Cancer Society (Other); NRG Oncology (Other)
Responsible Party: Principal Investigator, Maaike Oonk, Principle Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2016-00601; NRG-GY024 (Other: NRG)
Record Dates: First submitted 2021-08-15; First posted 2021-10-13 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Vulvar Cancer; Sentinel Lymph Node; Lymph Node Metastases
MeSH Terms: conditions — Vulvar Neoplasms; Lymphatic Metastasis | interventions — Cisplatin; Drug Therapy

STUDY DESIGN:
Intervention Model Description: phase II treatment trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chemoradiation (Experimental): Inguinofemoral radiotherapy (48-50 Gy in 1.8 Gy daily fractions, with a boost dose to the involved inguinal site for a total equivalent dose of 56 Gy over 5-6 weeks, preferably with simultaneous integrated boost technique) combined with weekly cisplatin 40 mg/m2 intravenously on days 1, 8, 15, 22 and 29
  Interventions: Radiation: Radiotherapy combined with cisplatin; Drug: Cisplatin

INTERVENTIONS:
Radiation: Radiotherapy combined with cisplatin — Inguinofemoral radiotherapy combined with weekly cisplatin
  Other Names: chemotherapy
Drug: Cisplatin — Inguinofemoral radiotherapy combined with weekly cisplatin

SUMMARY:
Vulvar cancer patients with SN-metastasis > 2mm will receive chemoradiation instead of an inguinofemoral lymphadenectomy.

DETAILED DESCRIPTION:
Rationale:

Standard treatment of early stage vulvar cancer is a wide local excision of the primary tumor combined with the sentinel node (SN) procedure for the groins. An inguinofemoral lymphadenectomy (IFL) is only indicated in case of a positive SN. An IFL is associated with major morbidity, e.g. wound healing problems, lymphoceles, lymphedema of the legs and recurrent infections. GROINSS-V II investigated whether radiotherapy would be a safe alternative for IFL in case of SN metastasis. The results for radiotherapy in the group with metastasis ≤ 2mm are promising. This study also showed that for metastasis > 2mm, only radiotherapy was not efficient. The efficacy of treatment can be increased by adding chemotherapy or giving a higher dose of radiotherapy. GROINSS-V III will investigate this regimen.

Objective:

The primary objective of this study is to investigate the safety of replacing inguinofemoral lymphadenectomy by chemoradiation in early stage vulvar cancer patients with a macrometastasis (>2mm) and/or extracapsular extension in the SN. The secondary objective is to evaluate the short and long-term morbidity associated with the SN procedure and chemoradiation.

Study design: Phase II treatment trial, with stopping rules for the incidence of groin recurrences.

Study population: early-stage vulvar cancer patients with a metastasis > 2mm in their SN, or more than one metastasis ≤ 2mm.

Intervention: Participants will be treated with chemoradiation, in a total dose of 56Gy to the involved site, combined with weekly cisplatin 40mg/m2

Main study parameters/endpoints: The primary endpoint is the groin recurrence rate in the first 2 years after primary treatment.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: participants will be treated with chemoradiation during 5 weeks instead of surgical treatment. There is a risk that this treatment will not be as effective as surgical treatment, which may lead to more groin recurrences which are hard to treat. By continuously monitoring the groin recurrence rate the investigators will notice activation of the stopping rule as early as possible.

ELIGIBILITY:
Inclusion Criteria:

* Histological confirmed primary SCC of the vulva
* T1 tumor, not encroaching urethra/vagina/anus
* Depth of invasion > 1mm
* Tumor diameter < 4cm
* Unifocal tumor
* No enlarged (>1.5cm) or suspicious inguinofemoral lymph nodes at imaging (CT/MRI/ultrasound)
* Possibility to obtain informed consent
* Metastatic sentinel lymph node; size of metastasis > 2mm and / or extracapsular extension, or
* Metastatic sentinel lymph node: more than 1 SN with metastasis ≤ 2mm
* Patients are able to understand requirements of study, provide written informed consent and comply with the study and follow-up procedures
* Adequate bone marrow, renal and liver function:

  * Absolute neutrophil count ≥ 1.5 x 109 /L
  * Platelet count ≥ 100 x 109 /L
  * Creatinine clearance ≥ 40 ml/min measured by the Cockroft Gault formula
  * Total bilirubin < 1.25 x ULN Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 2.5 x ULN
* Performance status of 0, 1 or 2 on the Eastern Cooperative Oncology Group (ECOG) Scale (Appendix A)
* Age 18 years or older
* Life expectancy of ≥ 12 weeks
* Written informed consent

Exclusion Criteria:

* Inoperable tumors and tumors > 4cm
* Multifocal tumors
* Tumors with other pathology than squamous cell carcinoma
* Patients with enlarged / suspicious lymph nodes which are proven metastatic after fine needle aspiration cytology
* No other carcinomas, other than basal cell carcinomas, within last 5 years
* History of pelvic radiotherapy
* History of any infection requiring hospitalization or antibiotics within 2 weeks before enrollment
* Pregnant female or nursing mother
* Desire to become pregnant
* Known brain or spinal cord metastases unless adequately treated (surgery or radiotherapy) with no evidence of progression and neurologically stable off anticonvulsants and steroids
* Unstable angina, myocardial infarction, cerebrovascular accident, > Class II congestive heart failure according to the New York Heart Association Classification for Congestive Heart Failure (see Appendix B) within 6 months before enrollment

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2028-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Groin recurrence rate | Within first 2 years after primary treatment
  Groin recurrence in the groin with SN metastasis treated with chemoradiation

SECONDARY OUTCOMES:
Treatment related morbidity | First two years after primary treatment
  Short and longterm morbidty
Quality of life as assessed using EORTC-QLQc30 | First two year after primary treatment
  Quality of life
Quality of life-vulvar cancer specific, as assessed using VU34 | First two year after primary treatment
  Quality of life-vulvar cancer specific

CONTACTS AND LOCATIONS:
Locations (27):
- United States (21):
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Mount Sinai Medical Center, Miami Beach, Florida
  - Baystate Medical Center, Springfield, Massachusetts
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Duke University Medical Center, Durham, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Women and Infants Hospital, Providence, Rhode Island
  - Avera Cancer Institute, Sioux Falls, South Dakota
- Netherlands (6):
  - Catharina Hospital Eindhoven, Eindhoven
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Radboud University Medical Center, Nijmegen
  - Erasmus Medical Center, Rotterdam
  - University Medical Center Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gien LT, Slomovitz B, Van der Zee A, Oonk M. Phase II activity trial of high-dose radiation and chemosensitization in patients with macrometastatic lymph node spread after sentinel node biopsy in vulvar cancer: GROningen INternational Study on Sentinel nodes in Vulvar cancer III (GROINSS-V III/NRG-GY024). Int J Gynecol Cancer. 2023 Apr 3;33(4):619-622. doi: 10.1136/ijgc-2022-004122. PMID 36653060